CLINICAL TRIAL: NCT04372602
Title: A Pilot Study of Duvelisib to Combat COVID-19
Brief Title: Duvelisib to Combat COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Verastem, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 202007009
Record Dates: First submitted 2020-04-30; First posted 2020-05-04 (Actual); Results first posted 2023-03-06 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: COVID-19
Keywords: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — duvelisib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Blocks of 10 patients will be used to allocate patients to duvelisib or placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Duvelisib (Experimental): -Duvelisib 25 mg twice daily for up to 10 days.
  Interventions: Drug: Duvelisib; Procedure: Peripheral blood draw
- Placebo (Sham Comparator): -Placebo 25 mg twice daily for up to 10 days.
  Interventions: Procedure: Peripheral blood draw; Drug: Placebo

INTERVENTIONS:
Drug: Duvelisib — -For patients unable to administer orally, a duvelisib suspension will be administered through a nasogastric/orogastric tube.
  Other Names: Copiktra
  Arms: Duvelisib
Procedure: Peripheral blood draw — * First 10 patients enrolled
  * Screening, Day 2, Day 4, Day 8, Day 10, Day 15, and Day 29
Drug: Placebo — -Provided by Verastem
  Arms: Placebo

SUMMARY:
The exceedingly high mortality rates of severe and critical COVID-19 warrant the identification and evaluation of novel therapies that could potentially mitigate the advanced disease manifestations. Based on preclinical data from this institution and others, the investigators hypothesize that PI3K inhibition with duvelisib could potentially quell aberrant hyperactivtation of the innate immune system, preferentially polarize macrophages, reduce pulmonary inflammation, and limit viral persistence, thereby improving patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of advanced COVID-19 as defined both of the following:

  * as a positive test for SARS-CoV-2 RNA detected by RT-PCR collected from the upper respiratory tract (e.g. nasopharyngeal, nasal, oropharyngeal swab, or saliva) and, if possible, the lower respiratory tract (sputum, tracheal aspirate, or bronchoalveolar lavage), analyzed by a CLIA certified lab with an FDA approved assay.
  * Critical disease manifested by any of the following:

    * Chest imaging with ≥ 50% lung involvement
    * Respiratory failure requiring invasive mechanical ventilation, non-invasive mechanical ventilation (eg. BiPAPA, OptiFlow), supplementary oxygen with FiO2 ≥ 6 LPM or extracorporeal membrane oxygenation (ECMO)
    * Shock - defined as mean arterial pressure ≤ 65 mmHg unresponsive to 25ml/kg isotonic intravenous fluid resuscitation and/or requiring vasopressor support
    * Cardiac dysfunction defined by:

      * New global systolic dysfunction with ejection fraction ≤ 40%
      * Takotsubo cardiomyopathy
* Patients who have received prior investigational or off-label agents for COVID-19 does not exclude eligibility.
* At least 18 years of age at the time of study registration
* Adequate hematologic function defined as absolute neutrophil count ≥1000/mm3 and platelet count ≥ 50,000/mm3 without growth factor or transfusion support for 7 days prior to screening.
* Creatinine-clearance ≥ 15 mL/minute or receiving renal replacement therapy
* Aminotransferase (AST/ALT) levels <3x the upper limit of normal
* Able to understand and willing to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable)
* Women of childbearing potential (defined as women with regular menses, women with amenorrhea, women with irregular cycles, women using a contraceptive method that precludes withdrawal bleeding, or women who have had a tubal ligation) are required to have a negative pregnancy test and use two forms of acceptable contraception, including one barrier method, during participation in the study treatment period.
* Male patients if engaging in sex with a women of childbearing potential are required to use two forms of acceptable contraception, including one barrier method, during participation in the study and throughout the evaluation period.

Exclusion Criteria:

* Known allergy or intolerance to duvelisib or another PI3K inhibitor.
* Known or suspected active viral (including CMV, HIV, hepatitis B, and hepatitis C), bacterial, mycobacterial, or fungal infection other than COVID-19. CMV viral load will be assessed at screening and those with viremia will be excluded. Other virologic testing not required unless infection is suspected.
* Pregnant and/or breastfeeding.
* Any uncontrolled intercurrent illness that would put the patient at greater risk or limit compliance with study requirements in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-10-12 (Actual); Primary Completion 2022-02-06 (Actual); Study Completion 2022-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John DiPersio, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goldsmith SR, Covut F, Fiala M, Xiang Z, Iqbal Z, Moore N, Bradtke E, Christen B, Rettig MP, Christ S, Gehrs L, Street E, Wallace N, Ritchey J, Gao F, Pachter J, Parikh B, Dubberke ER, DiPersio JF. Duvelisib for Critically Ill Patients With Coronavirus Disease 2019: An Investigator-Initiated, Randomized, Placebo-Controlled, Double-Blind Pilot Trial. Open Forum Infect Dis. 2023 Oct 27;10(11):ofad518. doi: 10.1093/ofid/ofad518. eCollection 2023 Nov. PMID 37953814
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Duvelisib | Placebo
Started | 15 | 13
Completed | 14 | 10
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Transitioned to comfort care | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Duvelisib | Placebo | Total
Number analyzed (Participants) | 15 | 13 | 28
Age, Continuous [Median (Full Range); unit: years] | 63 [26 to 79] | 64 [45 to 74] | 63 [26 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 9 | 8 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 13 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 5 | 11
  White | 9 | 8 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 13 | 28

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival as Measured by Number of Participants Alive Through 28 Days
Time Frame: Through 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Duvelisib | Placebo
Number analyzed (Participants) | 15 | 13
Participants | 10 | 8

2. Secondary Outcome: Length of Hospital Stay
Time Frame: Through 28 days
Measure: Median (Full Range); unit: days
Arm/Group | Duvelisib | Placebo
Number analyzed (Participants) | 15 | 13
days | 19 [7 to 28] | 24 [7 to 28]

3. Secondary Outcome: Length of ICU Stay
Time Frame: Through 28 days
Population: 1 participant was not evaluable in the placebo arm as the participant was not in the ICU.
Measure: Median (Full Range); unit: days
Arm/Group | Duvelisib | Placebo
Number analyzed (Participants) | 15 | 12
days | 19 [5 to 28] | 20.50 [7 to 28]

4. Secondary Outcome: Duration of Ventilator Use
Description: -For those on a ventilator at the time of randomization
Time Frame: Through 28 days
Population: 6 participants were not evaluable in the duvelisib arm as the participants were not on ventilators. 4 participants were not evaluable in the placebo arm as the participants were not on ventilators.
Measure: Median (Full Range); unit: days
Arm/Group | Duvelisib | Placebo
Number analyzed (Participants) | 9 | 9
days | 16 [2 to 28] | 20 [11 to 28]

5. Secondary Outcome: Duration of Vasopressors Use
Time Frame: Through 28 days
Population: 12 participants were not evaluable in the duvelisib arm as the participants did not receive vasopressors. 8 participants were not evaluable in the placebo arm as the participants did not receive vasopressors.
Measure: Median (Full Range); unit: days
Arm/Group | Duvelisib | Placebo
Number analyzed (Participants) | 3 | 5
days | 9 [7 to 28] | 19 [9 to 28]

6. Secondary Outcome: Duration on Renal Replacement Therapy
Time Frame: Through 28 days
Population: 14 participants were not evaluable in the duvelisib arm as the participants did not receive renal replacement therapy. 9 participants were not evaluable in the placebo arm as the participants did not receive renal replacement therapy.
Measure: Median (Full Range); unit: days
Arm/Group | Duvelisib | Placebo
Number analyzed (Participants) | 1 | 4
days | 28 [28 to 28] | 19 [13 to 28]

7. Secondary Outcome: Viral Kinetics as Measured by Virologic Failure
Description: -Defined as increase in viral load of >0.5 log on two consecutive days, or >1 log increase in one day, not in keeping with any baseline trend of rising viral loads during the pre-treatment viral testing
Time Frame: Through 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Duvelisib | Placebo
Number analyzed (Participants) | 15 | 13
Participants | 3 | 5

8. Secondary Outcome: Number of Adverse Events as Measured by CTCAE v. 5.0
Time Frame: Through 29 days
Measure: Count of Participants; unit: Participants
Arm/Group | Duvelisib | Placebo
Number analyzed (Participants) | 15 | 13
Participants
  Grade 1/2 anemia | 1 | 1
  Grade 3/4/5 anemia | 1 | 2
  Grade 1/2 leukocytosis | 0 | 1
  Grade 1/2 atrial fibrillation | 1 | 2
  Grade 3/4/5 cardiac arrest | 1 | 0
  Grade 1/2 pericarditis | 1 | 0
  Grade 1/2 sinus bradycardia | 1 | 1
  Grade 1/2 sinus tachycardia | 2 | 2
  Grade 1/2 ventricular arrhythmia | 0 | 1
  Grade 1/2 middle ear inflammation | 1 | 0
  Grade 1/2 conjunctivitis | 1 | 0
  Grade 3/4/5 corneal ulcer | 0 | 1
  Grade 3/4/5 colitis | 1 | 0
  Grade 1/2 constipation | 1 | 1
  Grade 1/2 diarrhea | 0 | 1
  Grade 3/4/5 gastroparesis | 1 | 0
  Grade 1/2 ileus | 2 | 0
  Grade 3/4/5 lower gastrointestinal hemorrhage | 1 | 1
  Grade 1/2 melena | 0 | 1
  Grade 3/4/5 mucositis oral | 1 | 0
  Grade 3/4/5 oral hemorrhage | 0 | 1
  Grade 3/4/5 pancreatitis | 1 | 0
  Grade 1/2 rectal ulcer | 0 | 1
  Grade 3/4/5 upper gastrointestinal hemorrhage | 0 | 1
  Grade 1/2 vomiting | 2 | 1
  Grade 3/4/5 vomiting | 1 | 1
  Grade 1/2 fever | 0 | 1
  Grade 3/4/5 fever | 0 | 1
  Grade 3/4/5 hypothermia | 0 | 1
  Grade 3/4/5 cholecystitis | 0 | 1
  Grade 1/2 bacteremia | 1 | 0
  Grade 3/4/5 conjunctivitis infective | 0 | 1
  Grade 1/2 lung infection | 0 | 1
  Grade 3/4/5 lung infection | 1 | 4
  Grade 3/4/5 sepsis | 1 | 2
  Grade 1/2 sinusitis | 1 | 0
  Grade 1/2 tracheitis | 0 | 1
  Grade 3/4/5 tracheitis | 0 | 1
  Grade 1/2 urinary tract infection | 0 | 1
  Grade 3/4/5 urinary tract infection | 0 | 1
  Grade 1/2 alanine aminotransferase increased | 2 | 2
  Grade 3/4/5 alkaline phosphatase increased | 0 | 1
  Grade 1/2 aspartate aminotransferase increased | 1 | 1
  Grade 1/2 blood bilirubin increased | 1 | 1
  Grade 1/2 elevated LFT NOS | 0 | 1
  Grade 1/2 platelet count decreased | 2 | 1
  Grade 1/2 acidosis | 1 | 0
  Grade 3/4/5 acidosis | 1 | 1
  Grade 1/2 hypercalcemia | 1 | 1
  Grade 1/2 hyperglycemia | 1 | 0
  Grade 1/2 hyperkalemia | 1 | 3
  Grade 3/4/5 hyperkalemia | 1 | 0
  Grade 1/2 hypernatremia | 2 | 1
  Grade 3/4/5 hypernatremia | 1 | 1
  Grade 1/2 hyperphosphatemia | 1 | 0
  Grade 1/2 hypoalbuminemia | 0 | 1
  Grade 1/2 hyponatremia | 2 | 0
  Grade 1/2 arthritis | 1 | 0
  Grade 3/4/5 intracranial hemorrhage | 1 | 1
  Grade 3/4/5 stroke | 1 | 0
  Grade 3/4/5 syncope | 1 | 0
  Grade 1/2 delirium | 0 | 1
  Grade 1/2 acute kidney injury | 1 | 0
  Grade 3/4/5 acute kidney injury | 1 | 0
  Grade 1/2 hematuria | 0 | 1
  Grade 3/4/5 hematuria | 1 | 2
  Grade 1/2 cough | 0 | 1
  Grade 1/2 epistaxis | 1 | 2
  Grade 3/4/5 epistaxis | 2 | 0
  Grade 3/4/5 hypoxia | 0 | 1
  Grade 3/4/5 pharyngeal hemorrhage | 1 | 1
  Grade 1/2 pneumothorax | 1 | 0
  Grade 3/4/5 respiratory failure | 6 | 5
  Grade 1/2 moisture associated skin damage | 1 | 0
  Grade 3/4/5 pressure ulcer | 0 | 1
  Grade 1/2 rash acneiform | 1 | 0
  Grade 1/2 skin tear | 1 | 1
  Grade 1/2 skin ulceration | 0 | 1
  Grade 3/4/5 subcutaneous emphysema | 1 | 0
  Grade 3/4/5 hematoma | 1 | 0
  Grade 1/2 hypotension | 2 | 2
  Grade 3/4/5 hypotension | 3 | 1
  Grade 3/4/5 peripheral ischemia | 0 | 1
  Grade 1/2 thromboembolic event | 0 | 1
  Grade 3/4/5 thromboembolic event | 1 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected from start of treatment through Day 29. All-cause mortality was collected from start of treatment through 6 months.
Arm/Group | Duvelisib | Placebo
All-Cause Mortality (participants affected / at risk) | 6/15 | 8/13
Serious Adverse Events (participants affected / at risk) | 6/15 | 8/13
Other Adverse Events (participants affected / at risk) | 15/15 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Duvelisib (N=15) | Placebo (N=13)
Cardiac arrest (Cardiac disorders) | 1 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Lung infection (Infections and infestations) | 1 | 2
Sepsis (Infections and infestations) | 0 | 1
Intracranial hemorrhage (Nervous system disorders) | 1 | 1
Stroke (Nervous system disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 | 5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Duvelisib (N=15) | Placebo (N=13)
Anemia (Blood and lymphatic system disorders) | 2 | 3
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 2
Pericarditis (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 1
Sinus tachycardia (Cardiac disorders) | 2 | 2
Ventricular arrhythmia (Cardiac disorders) | 0 | 1
Middle ear inflammation (Ear and labyrinth disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 0
Corneal ulcer (Eye disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Gastroparesis (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 2 | 0
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 1
Melena (Gastrointestinal disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 1 | 0
Oral hemorrhage (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Rectal ulcer (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 2
Fever (General disorders) | 0 | 2
Hypothermia (General disorders) | 0 | 1
Bacteremia (Infections and infestations) | 1 | 0
Conjunctivitis infective (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 3
Sepsis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Tracheitis (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 2
Alanine aminotransferase increased (Investigations) | 2 | 2
Alkaline phosphatase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1
Blood bilirubin increased (Investigations) | 1 | 1
Elevated LFT NOS (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 2 | 1
Acidosis (Metabolism and nutrition disorders) | 2 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 3 | 2
Hypernatremia (Metabolism and nutrition disorders) | 2 | 3
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 2
Hematuria (Renal and urinary disorders) | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Moisture associated skin damage (Skin and subcutaneous tissue disorders) | 1 | 0
Pressure ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 0
Skin tear (Skin and subcutaneous tissue disorders) | 1 | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 1
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 | 0
Hematoma (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 5 | 3
Peripheral ischemia (Vascular disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-30): https://cdn.clinicaltrials.gov/large-docs/02/NCT04372602/Prot_SAP_001.pdf